CLINICAL TRIAL: NCT02526524
Title: Randomized, Double-Blind, Parallel-Group, Multicenter, Placebo-Controlled, Dose-Ranging Study to Evaluate the Glycemic Effects, Safety, and Tolerability of Metformin Delayed Release In Subjects With Type 2 Diabetes Mellitus
Brief Title: Dose-Ranging Study to Evaluate the Glycemic Effects, Safety, and Tolerability of Metformin Delayed Release in Subjects With T2DM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elcelyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LCRM112
Record Dates: First submitted 2015-08-16; First posted 2015-08-18 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- 600 mg Met DR qAM (Experimental): 600 mg metformin delayed-release once daily in the morning
  Interventions: Drug: Met DR
- 900 mg Met DR qAM (Experimental): 900 mg metformin delayed-release once daily in the morning
  Interventions: Drug: Met DR
- 1200 mg Met DR qAM (Experimental): 1200 mg metformin delayed-release once daily in the morning
  Interventions: Drug: Met DR
- 1500 mg Met DR qAM (Experimental): 1500 mg metformin delayed-release once daily in the morning
  Interventions: Drug: Met DR
- Placebo-1 (Placebo Comparator): placebo match for 600 and 1200 mg Met DR qAM treatment groups
  Interventions: Drug: Placebo
- Placebo-2 (Placebo Comparator): placebo match for 900 and 1500 mg Met DR qAM treatment groups
  Interventions: Drug: Placebo
- 2000 mg Met IR (Active Comparator): 1000 mg metformin immediate-release twice daily
  Interventions: Drug: Met IR

INTERVENTIONS:
Drug: Met DR — metformin delayed-release tablets
  Arms: 1200 mg Met DR qAM; 1500 mg Met DR qAM; 600 mg Met DR qAM; 900 mg Met DR qAM
Drug: Met IR — metformin immediate-release tablets
  Arms: 2000 mg Met IR
Drug: Placebo
  Arms: Placebo-1; Placebo-2

SUMMARY:
The purpose of the study is to compare the glycemic effects of delayed-release metformin (Met DR) to placebo in subjects with type 2 diabetes mellitus (T2DM) over 16 weeks. The study is designed to evaluate several doses of Met DR (600 to 1500 mg once daily in the morning [qAM]) compared to placebo. A single-blind reference treatment of 2000 mg metformin immediate-release (Met IR) per day administered as equal divided doses (1000 mg Met IR BID) will also be included.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 25 years old at Visit 1 (Screening).
2. Is male, or is female and meets all of the following criteria:

   1. Not breastfeeding
   2. Negative pregnancy test result at Visit 1 (not applicable to post-menopausal or surgically sterile females)
   3. Surgically sterile, postmenopausal, or if of childbearing potential, must practice and be willing to continue to practice appropriate birth control during the entire duration of the study.
3. Body mass index (BMI) 20.0 to 45.0 kg/m² (inclusive) at Visit 1 (Screening).
4. Has a physical examination with no clinically significant abnormalities as judged by the investigator.
5. Has T2DM and an HbA1c of 7.5% to 10.5%, inclusive, at Visit 1.
6. Has an estimated glomerular filtration rate (eGFR) value of ≥60 mL/min/1.73 m² based on the Modification of Diet in Renal Disease (MDRD) equation.
7. Either is not treated with or has been on a stable treatment regimen with any of the following medications for a minimum of 3 months prior to Visit 1:

   1. Thiazolidinedione, sulfonylurea, dipeptidyl peptidase-4 inhibitors, and alpha-glucosidase inhibitors
   2. Hormone replacement therapy (female subjects) and testosterone (male subjects)
   3. Oral contraceptives (female subjects)
   4. Antihypertensive agents
   5. Lipid-lowering agents
   6. Thyroid replacement therapy
   7. Antidepressant agents
8. Ability to understand and willingness to adhere to protocol requirements.

Exclusion Criteria:

1. Has a clinically significant medical condition as judged by the investigator that could potentially affect study participation and/or personal well-being, including but not limited to the following conditions:

   1. Hepatic disease
   2. Gastrointestinal disease
   3. Endocrine disorder (T2DM is allowed)
   4. Cardiovascular disease
   5. Central nervous system diseases
   6. Psychiatric or neurological disorders
   7. Organ transplantation
   8. Chronic or acute infection
   9. Orthostatic hypotension, fainting spells or blackouts
   10. Allergy or hypersensitivity.
2. A history of diabetic ketoacidosis or hyperosmolar non-ketotic hyperglycemia within the past year.
3. Prior major surgery of any kind within 6 months of Visit 1.
4. A history of >3% weight change within 3 months of Visit 1.
5. A clinical laboratory test (clinical chemistry, hematology, or urinalysis) abnormality, other than that related to T2DM, judged by the investigator to be clinically significant at Visit 1.
6. An alanine aminotransferase or aspartate aminotransferase result >2.5 × upper limit of normal (ULN) or a bilirubin result >1.5 × ULN.
7. A physical, psychological, or historical finding that, in the investigator's opinion, would make the subject unsuitable for the study.
8. Has been treated, is currently being treated, or is expected to require or undergo treatment with any of the following excluded medications:

   1. Metformin within 2 months of Visit 1 (Screening)
   2. Insulin within 2 weeks of Visit 1 (Screening) or for more than 1 week within 3 months of Visit 1 (Screening)
   3. Glucagon-like peptide-1 receptor agonists or sodium-glucose co-transporter 2 inhibitors within 3 months of Visit 1
   4. Drugs known to affect body weight, including prescription medications and over-the-counter anti obesity agents within 3 months of Visit 1.
   5. Systemic corticosteroids by oral, intravenous, or intramuscular route; or potent, inhaled, or intrapulmonary steroids known to have a high rate of systemic absorption within 3 months of Visit 1
   6. Planned use of any drug treatment that affects gastric pH (prescription or over-the-counter), such as H2-receptor antagonists and proton pump inhibitors, after Visit 2 (Week -2), or planned chronic use of any antacids (i.e., more than twice per week) after Visit 2 (Week -2)
   7. Cationic drugs that are eliminated by renal tubular secretion within 1 week of Visit 1.
   8. Iodinated contrast dye within 1 week prior to Visit 1.
   9. Investigational drug within 2 months (or five half-lives of the investigational drug, whichever is greater) of the date of the first dose of randomized study medication.
   10. Met DR or double-blind matching placebo for Met DR at any time prior to Visit 1 (Screening)
9. Currently abuses drugs or alcohol or has a history of abuse that in the investigator's opinion would cause the individual to be noncompliant with study procedures.
10. Had a blood transfusion or experienced significant blood loss (i.e., >500 mL), including loss due to blood donation, within 2 months prior to Visit 1 (Screening), or is planning to donate blood during the study.
11. Has known immune system based allergies or hypersensitivity to any component of study treatment. A history of gastrointestinal intolerance to metformin is not exclusionary.
12. Is employed by Elcelyx Therapeutics, Inc. (that is an employee, contract worker, or designee of the company).
13. Has a fasting plasma glucose value >270 mg/dL at Visit 1 (Screening), Visit 2 (Week -2), and an unscheduled visit to be completed within 1 week following Visit 2. The unscheduled visit is to be completed only for subjects with a fasting plasma glucose value >270 mg/dL at Visit 1 and Visit 2.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Frias, MD, Principal Investigator — National Research Institute - Wilshire
Locations (137):
- United States (134):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Central Alabama Research, Birmingham, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Terence T. Hart, MD, Tuscumbia, Alabama
  - Radiant Research - Phoenix, Chandler, Arizona
  - Arrowhead Health Centers, Glendale, Arizona
  - Holland Center for Family Health, LTD, Peoria, Arizona
  - Elite Clinical Studies, Phoenix, Arizona
  - Thunderbird Internal Medicine - Indian School Rd., Phoenix, Arizona
  - Clinical Research Institute of Arizona, LLC, Surprise, Arizona
  - Summit Clinical Trials Center, Fayetteville, Arkansas
  - Searcy Medical Center, Searcy, Arkansas
  - Advanced Metabolic Care & Research Institute (AMCR), Escondido, California
  - MD Studies, Inc., Fountain Valley, California
  - National Research Institute, Huntington Park, California
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - Clinical Trials Research, Lincoln, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - National Research Institute, Los Angeles, California
  - Catalina Research Institute, Montclair, California
  - SRSD, Inc. dba Synergy San Diego, National City, California
  - Providence Clinical Research, North Hollywood, California
  - Pacific Research Partners, LLC, Oakland, California
  - SDS Clinical Trials, Inc., Orange, California
  - Center for Clinical Trials of Sacramento, Sacramento, California
  - Center for Clinical Trials of Scaramento, Sacramento, California
  - Superior Research LLC, Sacramento, California
  - Syrentis Clinical Research (formerly Research Across America), Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - Clinical Trial Investigators, Tustin, California
  - Infosphere Clinical Research, Van Nuys, California
  - Colorado Springs Health Partners, Colorado Springs, Colorado
  - Creekside Endocrine Associates, Denver, Colorado
  - Meridien Research - Brooksville, Brooksville, Florida
  - ALL Medical Research, LLC, Cooper City, Florida
  - Neostart Corporation dba AGA Clinical Trials, Hialeah, Florida
  - Care Partners Clinical Research, Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Family Health Care Clinical Studies, Kissimmee, Florida
  - Clinical Research of Central Florida-Lakeland, Lakeland, Florida
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - Tellus Clinical Research, Inc., Miami, Florida
  - Internal Research Associates LLC - Breton, Miami, Florida
  - Clinical Neuroscience Solutions, Inc. Healthcare Orlando, Orlando, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Private Practice - Andres Patron, DO, Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Meridien Reserach - St. Petersburg, St. Petersburg, Florida
  - Clinical Reserch Trials of Florida, Tampa, Florida
  - Meridien Research - Tampa, Tampa, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Biofortis, Inc., Addison, Illinois
  - AMR Sakeena Research, Aurora, Illinois
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Evanston Premier Healthcare Research LLC, Evanston, Illinois
  - Buynak Clinical Research, PC, Valparaiso, Indiana
  - The Iowa Clinic; Cardiovascular Services, West Des Moines, Iowa
  - Heartland Research Associates, LLC - Augusta, Augusta, Kansas
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - Otrimed, Edgewood, Kentucky
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - Louisville Metabolic and Atherosclerosis Research Center (L-MARC), Louisville, Kentucky
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Avant Research Associates, Crowley, Louisiana
  - Centex Studies, Inc. - lake Charles, Lake Charles, Louisiana
  - Columbia Medical Practice, Columbia, Maryland
  - Medstar Health Research Institute, Hyattsville, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Beacon Clinical Research, Quincy, Massachusetts
  - Radiant Research - Edina, Edina, Minnesota
  - Planters Clinic, Port Gibson, Mississippi
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Heartland Clinical Research, Omaha, Nebraska
  - Alliance Against Diabetes, Las Vegas, Nevada
  - AB Clinical Trials, Las Vegas, Nevada
  - Palm Medical Research, Las Vegas, Nevada
  - Ingham Neuroscience Group, LLC, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - NY Scientific, Brooklyn, New York
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - Mid-Hudson Medical Research, PLLC, Hopewell Junction, New York
  - Great Lakes Medical Research, Westfield, New York
  - PharmQuest, Greensboro, North Carolina
  - Triad Clinical Trials LLC, Greensboro, North Carolina
  - PMG Research of Rocky Mount, Rocky Mount, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Sterling Research Group, Ltd, Cincinnati, Ohio
  - Metabolic Atherosclerosis Research Center, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Urgent Care Specialists, LLC DBA Hometown Urgent Care and Occupational Health, Columbus, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Hometown Urgent Care and Research - Huber Heights, Huber Heights, Ohio
  - RAS Health LTD, Marion, Ohio
  - Summit Reserach Group, LLC, Stow, Ohio
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Medical Research South, LLC, Charleston, South Carolina
  - Mountain View Clinical Research - Greer, Greer, South Carolina
  - PMG of Charleston, LLC, Mt. Pleasant, South Carolina
  - Family Medicine of SayeBrook, LLC, Myrtle Beach, South Carolina
  - Hillcrest Clinical Research, LLC, Simpsonville, South Carolina
  - Palmetto Proactive Healthcare, LLC, Spartanburg, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - PMG Research of Bristol, LC - State, Bristol, Tennessee
  - PMG Research of Knoxville, Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Inc. - Memphis, Memphis, Tennessee
  - Trinity Clinical Research, Tullahoma, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - Trinity Universal Research Associates, Inc., Carrollton, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Galenos Research, Dallas, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Clinical Trial Network - Houston, Houston, Texas
  - Juno Research, LLC-Houston, Houston, Texas
  - Juno Research, LLC-Katy, Katy, Texas
  - Texas Diabetes Institute Research Center, San Antonio, Texas
  - Sun Research Institute, San Antonio, Texas
  - Victorium Clinical Research, San Antonio, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Southwest Health Associates, P.A., Sugar Land, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Burke Internal Medicine & Research, Burke, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Universal Research Group, LLC, Tacoma, Washington
- Puerto Rico (3):
  - Puerto Rico Renal and Health Research, Inc., Carolina
  - Advanced Medical Concepts, Cidra
  - Manati Center for Clinical Reserach Doctor's Center Hospital, Manatí

REFERENCES:
- [Derived] Henry RR, Frias JP, Walsh B, Skare S, Hemming J, Burns C, Bicsak TA, Baron A, Fineman M. Improved glycemic control with minimal systemic metformin exposure: Effects of Metformin Delayed-Release (Metformin DR) targeting the lower bowel over 16 weeks in a randomized trial in subjects with type 2 diabetes. PLoS One. 2018 Sep 25;13(9):e0203946. doi: 10.1371/journal.pone.0203946. eCollection 2018. PMID 30252913

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo match for 600 and 1200 mg Met DR qAM treatment groups (Placebo 1) and placebo match for 900 and 1500 mg Met DR qAM treatment groups (Placebo 2)
  Placebo
Period: Overall Study
Arm/Group | 600 mg Met DR qAM | 900 mg Met DR qAM | 1200 mg Met DR qAM | 1500 mg Met DR qAM | Placebo | 2000 mg Met IR
Started | 94 | 95 | 96 | 96 | 96 | 94
Completed | 82 | 86 | 70 | 89 | 72 | 73
Not Completed | 12 | 9 | 26 | 7 | 24 | 21
Not completed — Withdrawal by Subject | 3 | 3 | 6 | 1 | 9 | 5
Not completed — Adverse Event | 3 | 2 | 4 | 2 | 6 | 8
Not completed — Lost to Follow-up | 2 | 3 | 8 | 1 | 2 | 5
Not completed — Protocol Violation | 3 | 1 | 5 | 3 | 4 | 3
Not completed — Loss of Glucose Control | 0 | 0 | 3 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Sponsor Decision | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population: Subjects who took at least one dose of randomized study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | 600 mg Met DR qAM | 900 mg Met DR qAM | 1200 mg Met DR qAM | 1500 mg Met DR qAM | Placebo | 2000 mg Met IR | Total
Number analyzed (Participants) | 94 | 95 | 96 | 96 | 96 | 94 | 571
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (10.2) | 55 (10.5) | 55 (11.1) | 55 (8.9) | 57 (11.0) | 57 (11.1) | 56 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 38 | 45 | 42 | 53 | 45 | 269
  Male | 48 | 57 | 51 | 54 | 43 | 49 | 302
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 44 | 41 | 42 | 37 | 45 | 245
  Not Hispanic or Latino | 58 | 51 | 55 | 54 | 59 | 49 | 326
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Asian | 3 | 6 | 3 | 3 | 5 | 2 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Black or African American | 14 | 7 | 23 | 19 | 17 | 8 | 88
  White | 75 | 82 | 70 | 73 | 72 | 82 | 454
  More than one race | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Body Weight [Mean (Standard Deviation); unit: kg] | 94 (19.9) | 89 (18.5) | 93 (20.9) | 95 (22.2) | 86 (17.1) | 89 (21.3) | 91 (20.2)
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 33 (5.1) | 32 (5.5) | 32 (5.9) | 33 (5.8) | 31 (5.1) | 32 (5.4) | 32 (5.5)
HbA1c [Mean (Standard Deviation); unit: %] | 8.6 (0.85) | 8.7 (0.82) | 8.7 (0.90) | 8.6 (0.94) | 8.6 (0.87) | 8.6 (0.92) | 8.6 (0.88)
HbA1c stratum [Count of Participants; unit: Participants]
  <8.5% | 45 | 45 | 46 | 46 | 45 | 45 | 272
  ≥8.5% | 49 | 50 | 50 | 50 | 51 | 49 | 299
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 204 (58.1) | 202 (45.3) | 205 (59.0) | 212 (53.5) | 204 (57.3) | 200 (50.3) | 205 (54.0)
Diabetes Duration [Mean (Standard Deviation); unit: years] | 6.6 (5.20) | 8.8 (8.01) | 7.3 (6.25) | 7.6 (5.99) | 8.3 (6.99) | 8.6 (7.13) | 7.9 (6.67)
Estimated Glomerular Filtration Rate [Mean (Standard Deviation); unit: mL/min/1.73m²] | 94.4 (19.05) | 94.5 (22.83) | 96.2 (24.48) | 95.9 (22.77) | 96.4 (27.42) | 96.2 (22.42) | 95.6 (23.22)
Estimated Glomerular Filtration Rate Subgroup [Count of Participants; unit: Participants]
  <90 mL/min/1.73m² | 42 | 46 | 36 | 42 | 42 | 43 | 251
  ≥90 mL/min/1.73m² | 52 | 49 | 60 | 54 | 54 | 51 | 320
Prior Metformin Use [Count of Participants; unit: Participants] | 40 | 47 | 40 | 49 | 54 | 47 | 277

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (%) at 16 Weeks
Time Frame: Baseline and 16 weeks after the first dose of study medication
Population: Modified Intent-to-Treat: Subjects who took ≥1 dose of randomized study medication and had ≥1 post-Baseline value for HbA1c collected ≤1 week after discontinuing study medication and prior to administration of any new anti-diabetic medication with timing and/or dosage that may have reasonably influenced any subsequent glycemic data collected.
Measure: Least Squares Mean (Standard Error); unit: % glycated haemoglobin
Arm/Group | 600 mg Met DR qAM | 900 mg Met DR qAM | 1200 mg Met DR qAM | 1500 mg Met DR qAM | Placebo | 2000 mg Met IR
Number analyzed (Participants) | 88 | 93 | 88 | 94 | 90 | 89
% glycated haemoglobin | -0.33 (0.129) | -0.40 (0.123) | -0.49 (0.129) | -0.62 (0.124) | -0.06 (0.131) | -1.10 (0.129)
Statistical Analysis 1: Comparison: 600 mg Met DR qAM vs Placebo; Test type: Superiority; p = 0.1449, Mixed Models Analysis; Included treatment, visit, and treatment-by-visit interaction as fixed effects, and HbA1c value at Baseline as a covariate; LS Mean = -0.27, 95% CI 2-sided [-0.63 to 0.09], Standard Error of Mean 0.184
Statistical Analysis 2: Comparison: 900 mg Met DR qAM vs Placebo; Test type: Superiority; p = 0.0643, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean = -0.33, 95% CI 2-sided [-0.69 to 0.02], Standard Error of Mean 0.180
Statistical Analysis 3: Comparison: 1200 mg Met DR qAM vs Placebo; Test type: Superiority; p = 0.0214, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Means = -0.42, 95% CI 2-sided [-0.79 to -0.06], Standard Error of Mean 0.184
Statistical Analysis 4: Comparison: 1500 mg Met DR qAM vs Placebo; Test type: Superiority; p = 0.0022, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean = -0.55, 95% CI 2-sided [-0.91 to -0.20], Standard Error of Mean 0.180
Statistical Analysis 5: Comparison: Placebo vs 2000 mg Met IR; Test type: Superiority; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean = -1.03, 95% CI 2-sided [-1.39 to -0.67], Standard Error of Mean 0.184

ADVERSE EVENTS:
Time Frame: 16 Weeks
Arm/Group | 600 mg Met DR qAM | 900 mg Met DR qAM | 1200 mg Met DR qAM | 1500 mg Met DR qAM | Placebo | 2000 mg Met IR
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/95 | 0/96 | 0/96 | 1/96 | 0/94
Serious Adverse Events (participants affected / at risk) | 1/94 | 0/95 | 4/96 | 1/96 | 4/96 | 1/94
Other Adverse Events (participants affected / at risk) | 19/94 | 24/95 | 19/96 | 20/96 | 17/96 | 23/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 600 mg Met DR qAM (N=94) | 900 mg Met DR qAM (N=95) | 1200 mg Met DR qAM (N=96) | 1500 mg Met DR qAM (N=96) | Placebo (N=96) | 2000 mg Met IR (N=94)
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 600 mg Met DR qAM (N=94) | 900 mg Met DR qAM (N=95) | 1200 mg Met DR qAM (N=96) | 1500 mg Met DR qAM (N=96) | Placebo (N=96) | 2000 mg Met IR (N=94)
Diarrhoea (Gastrointestinal disorders) | 7 | 7 | 11 | 11 | 0 | 13
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 10 | 7 | 8 | 10 | 5
Nausea (Gastrointestinal disorders) | 3 | 3 | 1 | 3 | 1 | 9
Upper respiratory tract infection (Infections and infestations) | 1 | 5 | 1 | 0 | 2 | 2
Worsening Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study may be published by INSTITUTE, however the publication shall not disclose any SPONSOR Confidential Information, the INSTITUTE shall send the SPONSOR a copy of any such proposed publication 90 days prior to submission for publication, the INSTITUTE, on request of the SPONSOR, shall delete any SPONSOR Confidential Information in the proposed publication, and the INSTITUTE shall, on the SPONSOR's request, delay submission while the SPONSOR files applications for patents.